CLINICAL TRIAL: NCT00252694
Title: Effects of Candesartan Cilexetil (Candesartan) on Diabetic Retinopathy in Type 2 Diabetic Patients With Retinopathy.
Brief Title: DIabetic Retinopathy Candesartan Trials
Acronym: DIRECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2453C00047; DIRECT; SH-AHM-0047
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Results first posted 2014-06-06 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-04

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes mellitus type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — candesartan; candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- candesartan (Experimental): candesartan cilexetil 32 mg once daily
  Interventions: Drug: candesartan
- placebo (No Intervention): control

INTERVENTIONS:
Drug: candesartan — 32 mg oral tablet
  Other Names: ATACAND
  Arms: candesartan

SUMMARY:
The primary objective is to determine whether candesartan, compared to placebo reduces the progression of diabetic retinopathy in normoalbuminuric type 2 diabetic patients with retinopathy.

The secondary objective is to determine whether candesartan, compared to placebo, reduces the incidence of clinically significant macular oedema (CSME) and/or proliferative diabetic retinopathy (PDR) and beneficially influences the rate change in urinary albumin excretion rate (UAER).

This study is part of the DIRECT Programme also including a primary prevention study of diabetic retinopathy in type 1 diabetes and a secondary prevention study in type 1 diabetes. The primary objective for all three pooled studies is to determine whether candesartan, compared to placebo, reduces the incidence of microalbuminuria in type 1 and type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 37 - 75 years with type 2 diabetes diagnosed at age of 36 years or thereafter.
* Duration of diabetes for > 1 year and < 20 years with stable diabetic therapy within last 6 months.
* Patients with untreated resting mean sitting SBP < 130 mmHg and mean sitting DBP < 85 or treated resting mean SBP < 160 mmHg and mean sitting DBP < 90 mmHg with retinal photograph grading level >20/10 up to < 47/47 (on ETDRS severity scale).

Exclusion Criteria:

* Patients with the following conditions are excluded from participation in the study:
* Cataract or media opacity of a degree which precludes taking gradable retinal photographs
* Angle closure glaucoma, which precludes pharmacological dilatation of the pupil
* History of or presence of proliferative retinopathy
* History or presence of clinical significant macular oedema (CSME)
* History or evidence of photocoagulation of the retina
* Other retinal conditions which may mask assessment, eg, retinal vein occlusion
* Positive micral dipstick test
* Presence of secondary diabetes
* Pregnant or lactating women or women of child bearing potential not practicing an adequate method of contraception
* Need of treatment with ACE-inhibitor
* Haemodynamically significant aortic or mitral valve stenosis
* Known renal artery stenosis or kidney transplantation
* Hypersensitivity to study drug
* Severe concomitant disease which may interfere with the assessment of the patient, eg, malignancy, as judged by the investigator

Ages: 37 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4717 (Actual)
Dates: Start 2001-08; Primary Completion 2008-02 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Atacand Medical Science Director, MD, Study Director — AstraZeneca

REFERENCES:
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786
- [Derived] Tillin T, Orchard T, Malm A, Fuller J, Chaturvedi N. The role of antihypertensive therapy in reducing vascular complications of type 2 diabetes. Findings from the DIabetic REtinopathy Candesartan Trials-Protect 2 study. J Hypertens. 2011 Jul;29(7):1457-62. doi: 10.1097/HJH.0b013e3283480db9. PMID 21602709
- [Derived] Sjolie AK, Klein R, Porta M, Orchard T, Fuller J, Parving HH, Bilous R, Aldington S, Chaturvedi N. Retinal microaneurysm count predicts progression and regression of diabetic retinopathy. Post-hoc results from the DIRECT Programme. Diabet Med. 2011 Mar;28(3):345-51. doi: 10.1111/j.1464-5491.2010.03210.x. PMID 21309844
- [Derived] Porta M, Hainer JW, Jansson SO, Malm A, Bilous R, Chaturvedi N, Fuller JH, Klein R, Orchard T, Parving HH, Sjolie AK; DIRECT Study Group. Exposure to candesartan during the first trimester of pregnancy in type 1 diabetes: experience from the placebo-controlled DIabetic REtinopathy Candesartan Trials. Diabetologia. 2011 Jun;54(6):1298-303. doi: 10.1007/s00125-010-2040-1. Epub 2011 Jan 12. PMID 21225239
- [Derived] Bilous R, Chaturvedi N, Sjolie AK, Fuller J, Klein R, Orchard T, Porta M, Parving HH. Effect of candesartan on microalbuminuria and albumin excretion rate in diabetes: three randomized trials. Ann Intern Med. 2009 Jul 7;151(1):11-20, W3-4. doi: 10.7326/0003-4819-151-1-200907070-00120. Epub 2009 May 18. PMID 19451554
- [Derived] Sjolie AK, Klein R, Porta M, Orchard T, Fuller J, Parving HH, Bilous R, Chaturvedi N; DIRECT Programme Study Group. Effect of candesartan on progression and regression of retinopathy in type 2 diabetes (DIRECT-Protect 2): a randomised placebo-controlled trial. Lancet. 2008 Oct 18;372(9647):1385-93. doi: 10.1016/S0140-6736(08)61411-7. Epub 2008 Sep 25. PMID 18823658
- See also: CSR-D2453C00047.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1912&filename=CSR-D2453C00047.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled in the DIRECT Programme 8 June 2001 and last subject completed the DIRECT Programme 16 April 2008 mainly in hospital based clinics. A total of 4717 patients enrolled into the programme of whom 1905 patients proceeded to randomization into Study 47.
Pre-assignment Details: The most common reason for not being randomized was that all eligibility criteria were not fulfilled, followed by withdrawn informed consent.
Groups:
- Placebo: Placebo Comparator
Period: Overall Study
Arm/Group | Candesartan | Placebo
Started | 951 | 954
Completed | 807 | 800
Not Completed | 144 | 154
Not completed — Withdrawal by Subject | 83 | 91
Not completed — Death | 36 | 34
Not completed — Mostly Lost to Follow Up | 8 | 13
Not completed — Patient Moving | 17 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Candesartan | Placebo | Total
Number analyzed (Participants) | 951 | 954 | 1905
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 809 | 808 | 1617
  >=65 years | 142 | 146 | 288
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (7.6) | 56.8 (7.9) | 56.8 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 485 | 472 | 957
  Male | 466 | 482 | 948
Region of Enrollment [Number; unit: participants]
  Russian Federation | 162 | 165 | 327
  Europe | 419 | 438 | 857
  Israel | 188 | 173 | 361
  South Africa | 182 | 178 | 360

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a 3-step or Greater Increase in Early Treatment of Diabetic Retinopathy Study (EDTRS) Severity Scale
Description: 3 steps were defined as either a 1-step change in one eye and a 2-step change in the other eye or as a 3-step change in one eye only. EDRTS is a scale with 11 steps (1-11). A generlized log-rank test was used to test difference between treatments.
Time Frame: From baseline to end of study, i.e. 5 years, with visits after a half year, one year and thereafter one visit per year.
Population: The population was the Intention To Treat population which includes all randomized patients with any post-randomization data.
Measure: Number; unit: Participants
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 951 | 954
Participants | 161 (0.045) | 182 (0.052)
Statistical Analysis 1: Comparison: Candesartan vs Placebo; Test type: Superiority or Other; p = 0.1994, Log Rank; Generalized; Hazard Ratio (HR) = 0.870, 95% CI 2-sided [0.704 to 1.076]

2. Secondary Outcome: Number of Participants With at Least a 3 Step Improvement or a Persistent 2-step Improvement in the ETDRS Severity Scale.
Description: 3 steps were defined as either a 1-step change in one eye and a 2-step change in the other eye or as a 3-step change in one eye only. EDRTS is a scale with 11 steps (1-11).
Time Frame: From baseline to end of study, i.e. 5 years.
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 951 | 954
Participants | 180 (0.054) | 136 (0.040)

3. Secondary Outcome: Number of Participants With Incident Clinically Significant Macular Edema (CSME) and/or Proliferative Diabetic Retinopathy (PDR).
Description: Clinically Significant Macular Edema (CSME) and Proliferative Diabetic Retinopathy (PDR) are diagnosed via retinal photographs.
Time Frame: From baseline to end of study, i.e. 5 years.
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 951 | 954
Participants | 192 (0.06) | 193 (0.06)

4. Secondary Outcome: Rate of Change in Urinary Albumin Excretion Rate (UAER).
Description: An estimate of the slope from fitting a linear regression of log(UAER) over time (post-randomisation, yearly assessments) for each patient.
Time Frame: From Baseline to end of study, i.e. 5 years.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: log (µg/min)/1000 year
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 951 | 954
log (µg/min)/1000 year | 656 [605 to 708] | 718 [666 to 770]

ADVERSE EVENTS:
Time Frame: During treatment.
Description: The population used was the Safety population which includes all patients who received at least 1 dose of randomized study drug and for whom any post-dose data were available.
Arm/Group | Candesartan | Placebo
Serious Adverse Events (participants affected / at risk) | 301/949 | 267/953
Other Adverse Events (participants affected / at risk) | 50/949 | 18/953
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Candesartan (N=949) | Placebo (N=953)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 19 | 18
Angina Pectoris (Cardiac disorders) | 17 | 10
Acute Myocardial Infarction (Cardiac disorders) | 7 | 14
Angina Unstable (Cardiac disorders) | 7 | 10
Coronary Artery Disease (Cardiac disorders) | 3 | 10
Atrial Fibrillation (Cardiac disorders) | 9 | 3
Myocardial Ischaemia (Cardiac disorders) | 6 | 6
Acute Coronary Syndrome (Cardiac disorders) | 1 | 4
Arteriosclerosis Coronary Artery (Cardiac disorders) | 4 | 0
Cardiac Failure Congestive (Cardiac disorders) | 2 | 4
Coronary Artery Stenosis (Cardiac disorders) | 0 | 3
Cardiac Failure (Cardiac disorders) | 0 | 2
Supraventricular Tachycardia (Cardiac disorders) | 2 | 1
Aortic Valve Incompetence (Cardiac disorders) | 1 | 0
Aortic Valve Stenosis (Cardiac disorders) | 1 | 1
Arrhythmia Supraventricular (Cardiac disorders) | 1 | 0
Atrial Flutter (Cardiac disorders) | 1 | 0
Atrioventricular Block Complete (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1
Cardiac Disorder (Cardiac disorders) | 0 | 1
Cardiogenic Shock (Cardiac disorders) | 1 | 0
Cardiovascular Disorder (Cardiac disorders) | 0 | 1
Congestive Cardiomyopathy (Cardiac disorders) | 1 | 1
Coronary Artery Insufficiency (Cardiac disorders) | 1 | 0
Coronary Artery Occlusion (Cardiac disorders) | 1 | 0
Intracardiac Thrombus (Cardiac disorders) | 0 | 1
Ischaemic Cardiomyopathy (Cardiac disorders) | 0 | 1
Left Ventricular Failure (Cardiac disorders) | 1 | 0
Mitral Valve Disease (Cardiac disorders) | 1 | 0
Mitral Valve Incompetence (Cardiac disorders) | 1 | 0
Nodal Arrhythmia (Cardiac disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 1 | 1
Ventricular Septal Defect (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 2
Tinnitus (Ear and labyrinth disorders) | 2 | 0
Vertigo Positional (Ear and labyrinth disorders) | 2 | 0
Deafness Neurosensory (Ear and labyrinth disorders) | 0 | 1
Sudden Hearing Loss (Ear and labyrinth disorders) | 0 | 1
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 0 | 1
Goitre (Endocrine disorders) | 0 | 2
Basedow's Disease (Endocrine disorders) | 1 | 0
Cushing's Syndrome (Endocrine disorders) | 0 | 1
Thyroid Neoplasm (Endocrine disorders) | 0 | 1
Thyroiditis Chronic (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 11 | 6
Angle Closure Glaucoma (Eye disorders) | 0 | 1
Eye Haemorrhage (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 0 | 1
Open Angle Glaucoma (Eye disorders) | 1 | 0
Optic Ischaemic Neuropathy (Eye disorders) | 0 | 1
Optic Nerve Cupping (Eye disorders) | 1 | 0
Retinal Artery Embolism (Eye disorders) | 0 | 1
Retinal Detachment (Eye disorders) | 1 | 1
Retinal Tear (Eye disorders) | 1 | 0
Retinal Vein Occlusion (Eye disorders) | 1 | 1
Uveitis (Eye disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Anal Fistula (Gastrointestinal disorders) | 2 | 0
Gastroduodenitis (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 2 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 2
Pancreatitis Acute (Gastrointestinal disorders) | 2 | 1
Abdominal Adhesions (Gastrointestinal disorders) | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1
Colonic Polyp (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Duodenal Polyp (Gastrointestinal disorders) | 0 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Epigastric Discomfort (Gastrointestinal disorders) | 1 | 0
Erosive Oesophagitis (Gastrointestinal disorders) | 1 | 0
Food Poisoning (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastrointestinal Hypomotility (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal Perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Oesophagitis Ulcerative (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 1
Sigmoiditis (Gastrointestinal disorders) | 1 | 0
Umbilical Hernia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest Pain (General disorders) | 11 | 6
Non-Cardiac Chest Pain (General disorders) | 3 | 1
Sudden Death (General disorders) | 2 | 3
Sudden Cardiac Death (General disorders) | 2 | 1
Cardiac Death (General disorders) | 0 | 1
Death (General disorders) | 1 | 1
Inflammation (General disorders) | 1 | 0
Mass (General disorders) | 0 | 1
Multi-Organ Failure (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 7 | 5
Cholecystitis (Hepatobiliary disorders) | 3 | 2
Cholangitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1
Gallbladder Perforation (Hepatobiliary disorders) | 1 | 0
Hepatic Cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatic Steatosis (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1
Sphincter Of Oddi Dysfunction (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 2
Cellulitis (Infections and infestations) | 2 | 7
Pneumonia (Infections and infestations) | 2 | 6
Postoperative Wound Infection (Infections and infestations) | 5 | 0
Bronchitis (Infections and infestations) | 2 | 4
Diabetic Foot Infection (Infections and infestations) | 1 | 4
Gastroenteritis (Infections and infestations) | 4 | 3
Osteomyelitis (Infections and infestations) | 2 | 3
Perianal Abscess (Infections and infestations) | 3 | 2
Urinary Tract Infection (Infections and infestations) | 2 | 3
Diabetic Gangrene (Infections and infestations) | 2 | 0
Diverticulitis (Infections and infestations) | 2 | 1
Gangrene (Infections and infestations) | 1 | 2
Hepatitis C (Infections and infestations) | 2 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 2
Urosepsis (Infections and infestations) | 1 | 2
Viral Infection (Infections and infestations) | 2 | 1
Abscess (Infections and infestations) | 1 | 0
Abscess Limb (Infections and infestations) | 0 | 1
Acute Tonsillitis (Infections and infestations) | 0 | 1
Bronchiectasis (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 1
Cholecystitis Infective (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 1
Epstein-Barr Virus Infection (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 1
Herpes Zoster Ophthalmic (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1
Lobar Pneumonia (Infections and infestations) | 0 | 1
Localised Infection (Infections and infestations) | 1 | 1
Muscle Abscess (Infections and infestations) | 0 | 1
Osteomyelitis Chronic (Infections and infestations) | 1 | 0
Otitis Externa (Infections and infestations) | 1 | 0
Otitis Media (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Pericarditis Infective (Infections and infestations) | 1 | 0
Perineal Abscess (Infections and infestations) | 1 | 0
Post Procedural Infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 1
Salpingitis (Infections and infestations) | 0 | 1
Scrotal Abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1
Subcutaneous Abscess (Infections and infestations) | 0 | 1
Toxic Shock Syndrome (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 1
Viral Labyrinthitis (Infections and infestations) | 1 | 0
Viral Pericarditis (Infections and infestations) | 0 | 1
Wound Infection (Infections and infestations) | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 3
Head Injury (Injury, poisoning and procedural complications) | 3 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 3 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 2 | 1
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 2
Limb Injury (Injury, poisoning and procedural complications) | 2 | 1
Meniscus Lesion (Injury, poisoning and procedural complications) | 2 | 0
Multiple Injuries (Injury, poisoning and procedural complications) | 1 | 2
Acetabulum Fracture (Injury, poisoning and procedural complications) | 1 | 0
Alcohol Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Asphyxia (Injury, poisoning and procedural complications) | 1 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Dislocation Of Joint Prosthesis (Injury, poisoning and procedural complications) | 1 | 0
Dural Tear (Injury, poisoning and procedural complications) | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 1
Forearm Fracture (Injury, poisoning and procedural complications) | 1 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 1
Internal Injury (Injury, poisoning and procedural complications) | 1 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0
Joint Injury (Injury, poisoning and procedural complications) | 0 | 1
Multiple Fractures (Injury, poisoning and procedural complications) | 1 | 0
Muscle Injury (Injury, poisoning and procedural complications) | 1 | 0
Peroneal Nerve Injury (Injury, poisoning and procedural complications) | 1 | 0
Poisoning (Injury, poisoning and procedural complications) | 0 | 1
Postoperative Hernia (Injury, poisoning and procedural complications) | 1 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1
Soft Tissue Injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 1
Sternal Fracture (Injury, poisoning and procedural complications) | 1 | 0
Tendon Injury (Injury, poisoning and procedural complications) | 1 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 1 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 1
Red Blood Cell Sedimentation Rate Increased (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 7
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 4 | 6
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 6
Diabetic Foot (Metabolism and nutrition disorders) | 2 | 4
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 0 | 3
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Chondrocalcinosis Pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1
Dupuytren's Contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Jaw Cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Trigger Finger (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 6
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adrenal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adrenal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign Gastrointestinal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Biliary Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gallbladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Glioblastoma Multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Kaposi's Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Squamous Cell Carcinoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases To Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myeloproliferative Disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nasal Cavity Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm Prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Peripheral T-Cell Lymphoma Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 10 | 9
Transient Ischaemic Attack (Nervous system disorders) | 1 | 6
Diabetic Neuropathy (Nervous system disorders) | 4 | 1
Syncope (Nervous system disorders) | 4 | 2
Carpal Tunnel Syndrome (Nervous system disorders) | 3 | 1
Cerebral Infarction (Nervous system disorders) | 1 | 3
Ischaemic Stroke (Nervous system disorders) | 3 | 1
Loss Of Consciousness (Nervous system disorders) | 2 | 0
Sciatica (Nervous system disorders) | 2 | 0
Vith Nerve Paralysis (Nervous system disorders) | 0 | 2
Vertebrobasilar Insufficiency (Nervous system disorders) | 2 | 0
Brain Stem Infarction (Nervous system disorders) | 1 | 0
Cerebral Ischaemia (Nervous system disorders) | 0 | 1
Diabetic Hyperosmolar Coma (Nervous system disorders) | 1 | 0
Diabetic Neuropathic Ulcer (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Embolic Stroke (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Facial Palsy (Nervous system disorders) | 1 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Ischaemic Cerebral Infarction (Nervous system disorders) | 1 | 0
Lumbar Spinal Stenosis (Nervous system disorders) | 1 | 0
Myasthenia Gravis (Nervous system disorders) | 0 | 1
Neuritis (Nervous system disorders) | 1 | 0
Neuritis Cranial (Nervous system disorders) | 1 | 0
Partial Seizures (Nervous system disorders) | 0 | 1
Radial Nerve Palsy (Nervous system disorders) | 0 | 1
Spondylitic Myelopathy (Nervous system disorders) | 0 | 1
Subarachnoid Haemorrhage (Nervous system disorders) | 0 | 1
Syncope Vasovagal (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Anxiety Disorder (Psychiatric disorders) | 0 | 1
Depression Suicidal (Psychiatric disorders) | 1 | 0
Generalised Anxiety Disorder (Psychiatric disorders) | 0 | 1
Major Depression (Psychiatric disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 3 | 1
Renal Colic (Renal and urinary disorders) | 0 | 3
Urinary Incontinence (Renal and urinary disorders) | 2 | 0
Bladder Prolapse (Renal and urinary disorders) | 0 | 1
Calculus Ureteric (Renal and urinary disorders) | 1 | 1
Calculus Urethral (Renal and urinary disorders) | 1 | 0
Calculus Urinary (Renal and urinary disorders) | 1 | 1
Cystocele (Renal and urinary disorders) | 1 | 1
Diabetic Nephropathy (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephropathy (Renal and urinary disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Stress Urinary Incontinence (Renal and urinary disorders) | 1 | 0
Ureteric Stenosis (Renal and urinary disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 1 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 2
Breast Mass (Reproductive system and breast disorders) | 1 | 0
Cervical Dysplasia (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Ovarian Cyst (Reproductive system and breast disorders) | 1 | 0
Pelvic Peritoneal Adhesions (Reproductive system and breast disorders) | 1 | 0
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Testicular Cyst (Reproductive system and breast disorders) | 0 | 1
Uterine Polyp (Reproductive system and breast disorders) | 1 | 0
Vaginal Prolapse (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 2
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic Neuropathic Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic Ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Lichen Planus (Skin and subcutaneous tissue disorders) | 1 | 0
Neuropathic Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Sebaceous Hyperplasia (Skin and subcutaneous tissue disorders) | 0 | 1
Femoral Artery Occlusion (Vascular disorders) | 0 | 3
Hypertension (Vascular disorders) | 3 | 1
Hypertensive Crisis (Vascular disorders) | 1 | 3
Aortic Arteriosclerosis (Vascular disorders) | 2 | 0
Arteriosclerosis (Vascular disorders) | 0 | 2
Peripheral Vascular Disorder (Vascular disorders) | 1 | 2
Aortic Stenosis (Vascular disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 1
Extremity Necrosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Ischaemia (Vascular disorders) | 0 | 1
Microangiopathy (Vascular disorders) | 1 | 0
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 | 1
Peripheral Ischaemia (Vascular disorders) | 1 | 0
Varicose Vein (Vascular disorders) | 0 | 1
Venous Thrombosis Limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Candesartan (N=949) | Placebo (N=953)
Hypotension (Vascular disorders) | 50 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No